CLINICAL TRIAL: NCT03724084
Title: A Phase 1b/2 Study of Pinometostat in Combination With Standard Induction Chemotherapy in Newly Diagnosed Acute Myeloid Leukemia With MLL Rearrangement
Brief Title: Pinometostat With Standard Chemotherapy in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia and MLL Gene Rearrangement
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Other - Study agent no longer available
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02349; NCI-2018-02349 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10212 (Other: Ohio State University Comprehensive Cancer Center LAO); 10212 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; EPZ-5676

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (higher and lowers dose pinometostat) (Experimental): Patients receive higher dose pinometostat IV continuously on days 1-7 and lower dose pinometostrat IV continuously on days 8-35. Patients also receive daunorubicin hydrochloride IV over 10-30 minutes on days 8-10 and cytarabine IV continuously on days 8-14. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve CR/CRi after treatment receive pinometostat IV continuously on days 1-28, daunorubicin hydrochloride IV over 10-30 minutes on days 1 and 2 and cytarabine IV continuously on days 1-5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Pinometostat
- Cohort II (higher dose pinometostat) (Experimental): Patients receive higher dose pinometostat intravenously (IV) continuously on days 1-35. Patients also receive daunorubicin hydrochloride IV over 10-30 minutes on days 8-10 and cytarabine IV continuously on days 8-14. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve CR/CRi after treatment receive pinometostat IV continuously on days 1-28, daunorubicin hydrochloride IV over 10-30 minutes on days 1 and 2 and cytarabine IV continuously on days 1-5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Pinometostat

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Pinometostat — Given IV
  Other Names: DOT1L Inhibitor EPZ-5676; EPZ-5676

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of pinometostat and how well it works with standard chemotherapy in treating patients with newly diagnosed acute myeloid leukemia and a type of genetic mutation called MLL gene rearrangement. Pinometostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in standard chemotherapy, such as daunorubicin hydrochloride and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pinometostat with standard chemotherapy may work better at treating acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine a safe and tolerable schedule of pinometostat continuous intravenous infusion in combination with daunorubicin hydrochloride (daunorubicin) and cytarabine in patients with untreated, newly diagnosed acute myeloid leukemia harboring MLL rearrangement.

II. Determine the rate of complete remission (complete remission [CR], CR with incomplete hematologic recovery [CRi]) in patients with newly diagnosed acute myeloid leukemia harboring MLL rearrangement after treatment with pinometostat in combination with daunorubicin and cytarabine.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. Estimate biologic activity of 7 day window treatment of pinometostat monotherapy.

III. Estimate the toxicity profile of pinometostat alone (week 1) and in combination with daunorubicin and cytarabine.

IV. Estimate event free and overall survival of patients with MLL rearranged acute myeloid leukemia after combination treatment with pinometostat, daunorubicin, and cytarabine.

V. Estimate the early death rate (death =< 30 days) of pinometostat, daunorubicin, and cytarabine.

VI. Determine the rate of minimal residual disease (MRD) negativity by clinical flow cytometry on post-treatment recovery bone marrow.

OUTLINE: This is a phase I, dose-escalation study of pinometostat followed by a phase II study. Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive higher dose pinometostat intravenously (IV) continuously on days 1-7 and lower dose pinometostrat IV continuously on days 8-35. Patients also receive daunorubicin hydrochloride IV over 10-30 minutes on days 8-10 and cytarabine IV continuously on days 8-14. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve CR/CRi after treatment receive pinometostat IV continuously on days 1-28, daunorubicin hydrochloride IV over 10-30 minutes on days 1 and 2 and cytarabine IV continuously on days 1-5 in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive higher dose pinometostat IV continuously on days 1-35. Patients also receive daunorubicin hydrochloride IV over 10-30 minutes on days 8-10 and cytarabine IV continuously on days 8-14. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve CR/CRi after treatment receive pinometostat IV continuously on days 1-28, daunorubicin hydrochloride IV over 10-30 minutes on days 1 and 2 and cytarabine IV continuously on days 1-5 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 1 year, then every 3 months for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed acute myeloid leukemia by World Health Organization (WHO) criteria. Patients with treatment-related acute leukemia are eligible if they do not exceed lifetime anthracycline doses
* Presence of a cytogenetic rearrangement of KMT2A (MLL) by interphase fluorescent in-situ hybridization (FISH)
* Patients must have previously untreated (with exception of hydroxyurea for count control or all-trans retinoic acid [ATRA] for acute promyelocytic leukemia [APML] that was initially suspected but later ruled out) AML by World Health Organization (WHO) criteria. Treatment with hydroxyurea for count-control of hyperproliferative disease is permitted before and during treatment with pinometostat and chemotherapy
* Age >=14 years at time of screening, although individual sites may further restrict age eligibility in accordance with local Institutional Review Board (IRB) and hospital policy.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), unless elevated due to Gilbert syndrome, hemolysis, or leukemia (at the time of eligibility screening)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN, unless due to leukemia in which case < 5 x ULN (at the time of eligibility screening)
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (at the time of eligibility screening)
* Glomerular filtration rate (GFR) => 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (both) (at the time of eligibility screening)
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial (at the time of eligibility screening)
* If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated (at the time of eligibility screening)
* If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load (at the time of eligibility screening)
* For pediatric patients, a serum creatinine based on age/gender as follows:

  * 10 to < 13 years: male = 1.2; female = 1.2
  * 13 to < 16 years: male = 1.3; female = 1.4
  * >= 16 years: male = 1.7; female = 1.4
* Be medically fit, in the opinion of the investigator, for intensive (7+3) induction chemotherapy
* Left ventricular ejection fraction (LVEF) >= 45% confirmed by echocardiogram or multi-gated acquisition scan (MUGA), AND no symptoms of congestive heart failure exceeding New York Heart Association (NYHA) class II
* Willingness to comply with all study procedures, including scheduled visits, investigational and standard of care drug administration plans, imaging studies, laboratory tests (including all biomarkers), procedures, and study- and disease-related restrictions
* The effects of pinometostat on the developing human fetus are unknown. For this reason and because other small molecule inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation, and for 4 weeks after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate barrier contraception prior to the study, for the duration of study participation, and for 90 days after completion of pinometostat administration
* Ability to understand and the willingness to sign a written informed consent document or, for patients with impaired decision-making capacity, the consent of a close legal guardian who is readily available

Exclusion Criteria:

* Acute promyelocytic leukemia with t(15;17)(q22;q12) and/or PML-RARA molecular rearrangement, or other atypical RARA translocation partner
* Patients who have received prior chemotherapy for AML, excluding hydroxyurea for count control, or ATRA for APML that was initially suspected but later ruled out
* Patients who have received any prior investigational agent for acute myeloid leukemia
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have a cumulative lifetime exposure (prior to study entry) of greater than 300 mg/m^2 doxorubicin equivalent anthracycline
* Patients who have received chest radiation (unless organ-sparing) and who have a cumulative lifetime exposure (prior to study entry) of greater than 240 mg/m^2 doxorubicin equivalent anthracycline
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia, or peripheral neuropathy (up to grade 2 is permitted)
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pinometostat or other agents used in study
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible unless the offending medication can be safely stopped prior to enrollment. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (with exception), symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia not controllable with medications, electrocardiographic evidence of ischemia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients receiving an anti-microbial agent may be eligible if the patient remains afebrile and hemodynamically stable for 72 hours
* Patients with an active bleeding diathesis
* Pregnant women are excluded from this study because pinometostat is a small molecule inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pinometostat, breastfeeding should be discontinued if the mother is treated with pinometostat. These potential risks may also apply to other agents used in this study
* Subjects with known symptomatic leukemia of the central nervous system including leptomeningeal leukemic involvement
* History of active other malignancy that limits survival to less than 1 year
* Ongoing viral or drug induced liver injury, including active chronic hepatitis C virus (HCV), chronic active hepatitis B, clinically known alcoholic liver disease, non-alcoholic steatohepatitis, non-alcoholic fatty liver disease, primary biliary cirrhosis, other cirrhosis of the liver, history of hepatic encephalopathy, or portal hypertension
* Any other prior condition that could, in the opinion of the investigator, compromise patient safety or evaluation of the primary outcome

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James S Blachly, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I (Higher and Lower Dose Pinometostat): Patients receive higher dose pinometostat IV continuously on days 1-7 and lower dose pinometostrat IV continuously on days 8-35. Patients also receive daunorubicin hydrochloride IV over 10-30 minutes on days 8-10 and cytarabine IV continuously on days 8-14. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve CR/CRi after treatment receive pinometostat IV continuously on days 1-28, daunorubicin hydrochloride IV over 10-30 minutes on days 1 and 2 and cytarabine IV continuously on days 1-5 in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (Phase Ib)
Description: Dose escalation for phase 1b will be in the usual 3+3 fashion
Time Frame: Up to 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

2. Primary Outcome: Complete Response (CR) or Complete Response With Incomplete Count Recovery (CRi) Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 3 | 3
participants | 3 | 2

3. Secondary Outcome: Number of Participants With Incidence of Adverse Events
Description: Will be graded and reported according to Common Terminology Criteria for Adverse Events version 5. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Time Frame: For up to 3 years
Measure: Number; unit: participants
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 3 | 3
participants
  Any grade | 3 | 3
  Grade 4 | 3 | 2

4. Secondary Outcome: Time to Hematologic Count Recovery
Description: Will be analyzed using lab evaluation of complete blood counts and differential.
Time Frame: Up to 3 years
Population: Data not collect and analyzed
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Differential Blast Counts
Description: Will be analyzed using lab evaluation of complete blood counts and differential.
Time Frame: Baseline up to day 8
Population: Data was not collected and analyzed
Arm/Group | Cohort I (Higher and Lowers Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Rate of Minimal Residual Disease (MRD) Positivity
Description: Will be evaluated by multiparameter flow cytometry, next-generation sequencing (or both) after induction therapy among those patients who attain morphologic and cytogenetic CR. Will be calculated with the exact binomial 95% confidence intervals.
Time Frame: Up to 3 years
Population: Data not collected and analyzed due to early study termination
Arm/Group | Cohort I (Higher and Lowers Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the start of study treatment until progression or death, whichever occurs earliest, assessed up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort I (Higher and Lowers Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 3 | 1
Days | 100 [95 to 133] | 400 [400 to 400]

8. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort I (Higher and Lowers Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
Number analyzed (Participants) | 3 | 2
Days | 326 [181 to 450] | 298 [168 to 428]

ADVERSE EVENTS:
Time Frame: The Adverse event information was collected for study patients from baseline through study completion utilizing the CTCAE version 5.0 to determine the severity of the reaction for adverse event reporting from baseline to after study completion, up to 2 years, All-Cause Mortality monitored/assessed up to 3 years.
Arm/Group | Cohort I (Higher and Lower Dose Pinometostat) | Cohort II (Higher Dose Pinometostat)
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Higher and Lower Dose Pinometostat) (N=3) | Cohort II (Higher Dose Pinometostat) (N=3)
White blood cell decreased (Investigations) | 3 (3) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Higher and Lower Dose Pinometostat) (N=3) | Cohort II (Higher Dose Pinometostat) (N=3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (14) | 1 (6)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (8) | 1 (2)
Platelet count decreased (Investigations) | 3 (22) | 2 (5)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
White blood cell decreased (Investigations) | 3 (11) | 1 (2)
INR increased (Investigations) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 2 (4)
Edema Limbs (General disorders) | 2 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated early due to investigational product not being available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03724084/Prot_SAP_000.pdf
  • Informed Consent Form: P10212_A01Consent(Redacted) (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03724084/ICF_001.pdf
  • Informed Consent Form: P10212_A01ConsentAssentForm(Redacted) (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03724084/ICF_002.pdf
  • Informed Consent Form: P10212_A01ConsentParentalPermission(Redacted) (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03724084/ICF_003.pdf